CLINICAL TRIAL: NCT00557622
Title: Clinical Evaluation of BRL29060A (Paroxetine Hydrochloride Hydrate) in Posttraumatic Stress Disorder (PTSD) - A Placebo-controlled, Single-Blind Comparative Study -
Brief Title: Clinical Evaluation of BRL29060A (Paroxetine Hydrochloride Hydrate) in Posttraumatic Stress Disorder (PTSD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: difficulty in achieving target enrollment numbers
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIR109164
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Results first posted 2009-11-19 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Post-Traumatic Stress Disorder; Stress Disorders, Post-Traumatic
Keywords: PTSD (Posttraumatic Stress Disorder); CAPS; fMRI; Paroxetine
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Paroxetine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- paroxetine (Experimental): Drug 2 (20 mg/day or placebo) will be administered once daily after supper for the first two weeks after the run-in phase. If the investigator/subinvestigator judges that a sufficient response is achieved, Drug 2 will be continued for the remaining period. If a sufficient response is not achieved with Drug 2 but treatment is well tolerated, the dose will be titrated to one step higher level until a sufficient response is achieved [i.e., Drug 3 (30 mg/day or placebo) → Drug 4 (40 mg/day or placebo) → Drug 5 (50 m/day or placebo)] at intervals of at least two weeks by once daily administration after supper. Once a sufficient response is achieved, that dose will be continued.
  Interventions: Drug: paroxetine
- placebo (Placebo Comparator): placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: paroxetine — BRL29060A (paroxetine hydrochloride hydrate, hereafter paroxetine) administered orally over the dose range of 20 mg to 50 mg once daily after supper for 12 weeks in Japanese patients with posttraumatic stress disorder (PTSD)
  Arms: paroxetine
Other: placebo — placebo
  Arms: placebo

SUMMARY:
This is a single-blind, placebo-controlled, parallel group study to evaluate the efficacy of BRL29060A (paroxetine hydrochloride hydrate, hereafter paroxetine) administered orally over the dose range of 20 mg to 50 mg once daily after supper for 12 weeks in Japanese patients with posttraumatic stress disorder (PTSD) as assessed by the change from baseline in CAPS-SX total score. Also the effect of paroxetine on regional cerebral blood flow (rCBF) induced by subthreshold emotional arousing (or symptom stimulating) tasks will be determined using functional magnetic resonance imaging (fMRI) for exploratory assessment of the correlation between the change in rCBF and the efficacy.

The sample size is 30 subjects. The study period consists of 4 weeks of run-in phase, 12 weeks of treatment phase, 0-3 weeks of taper phase and follow-up examination at 2 weeks after the last dose, for a total of 18-21 weeks.

Subjects will visit the clinic at the start of run-in phase, Week -2, the start of treatment phase, Weeks 2, 4, 6, 8 and 12 of treatment, and follow-up examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are primarily diagnosed with PTSD (Posttraumatic Stress Disorder: 309.81) using DSM-IV-TR criteria. The CAPS-DX (Clinician-Administered PTSD Scale-DX) and M.I.N.I. (The Mini International Neuropsychiatric Interview, Japanese version 5.0.0. [2003]) will be used for diagnosis
* Pathologic condition: Patients who experienced a motor vehicle accident (MVA) with severe or potential severe physical injury more than 3 months ago but less than 12 months ago
* Patients aged 20 and <65 at the time of signing the Informed consent
* Male and female patients
* Inpatient/outpatient status: Both are permitted
* Patients who are able to give written informed consent in person (i.e., patients who are capable of giving written informed consent on their own)
* Patients whose combined score of the CAPS-SX standard B, C, and D is over 50

Exclusion Criteria:

* Patients primarily diagnosed with a DSM-IV-TR Axis I disorder other than PTSD (e.g. major depressive disorder, dysthymic disorder, specific phobia [simple phobia], obsessive-compulsive disorder, panic disorder, etc.) within 6 months of week -4 (start of baseline phase)
* Patients presenting with a current major depressive episode that preceded the diagnosis of PTSD
* Patients receiving disability payments due to PTSD or other psychiatric diseases
* Patients currently engaged in compensation litigation whereby personal gain would be achieved from prolonged symptoms of PTSD or any other psychiatric disorders
* Patients who meet the DSM-IV-TR criteria for substance abuse or dependence (alcohol or drugs) within 6 months of Week -4 (start of baseline phase)
* Patients with history of a suicide attempt within 6 months before Week -4 (start of baseline phase), or have, in the opinion of the investigator, "C. high risk of suicide" according to the MINI at Week -4
* Patients who are pregnant, lactating or of childbearing potential and are likely to become pregnant
* Patients receiving electro-convulsive therapy (ECT) prior to Week -4 (start of baseline phase)
* Patients receiving another investigational product within 12 weeks before Week -4 (start of baseline phase)
* Patients with a history or complication of manic psychosis
* Patients with a history or complication of convulsive disorder (epilepsy, etc.)
* Patients with a diagnosis or complication of a cognitive disorder (MMSE <=24 points)
* Patients with a history and complication of serious cerebral organic disorder. (e.g. cerebrovascular disorder, meningitis, degenerative disease and other neurological disorders and seizures; however, bleeding in the upper arachnoid membrane should not be excluded)
* Patients unable or unwilling to undergo the fMRI procedure (e.g., cerebrovascular clipping surgery, pacemaker, any internal metals with magnetism, and claustrophobia)
* Patients with glaucoma
* Patients with a known tendency for bleeding or those with predisposing conditions
* Patients with a history of hypersensitivity to paroxetine
* Patients with serious physical symptoms (cardiac, hepatic and renal dysfunction, or hematopoietic dysfunction, etc.). For seriousness, Grade 3 of "Criteria for seriousness of adverse reactions to drugs, etc. (Yakuan No.80)" is used as an index
* Patients with a history or complication of cancer or malignant tumour
* Patients with chronic hepatitis type B and/or C which is positive of hepatitis B surface antigen (HBsAg) and/or hepatitis C antibody
* Others whom the investigator or sub-investigator considers ineligible for or unable to participate in the investigation
* Criteria at Week 0 (start of Treatment Phase):

Subjects whose drug compliance rate for Drug 1 (Run-in Phase placebo) is <80% between Week -4 and Week 0;

Subjects whose CAPS-SX total score of the standard B, C, and D at Week 0 varied by 25% or more compared with those at Week -2

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-01-25 (Actual); Primary Completion 2008-12-11 (Actual); Study Completion 2008-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Japan (2):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Tokyo

REFERENCES:
- [Background] This study has not been published in the scientific literature.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to assignment to the 12-week treatment phase, all participants received placebo in a single-blind manner in a 4-week run-in phase. Participants completing the run-in phase were then randomized to receive either placebo or paroxetine for the remainder of the study. Two participants were withdrawn from the study before randomization.
Groups:
- Placebo: Placebo once daily (OD)
- Paroxetine 20-50 mg/Day: Paroxetine 20 milligrams (mg)/day once daily (OD) for 2 weeks; titration up to 50 mg/day OD if necessary to achieve sufficient response. The last dose level in the treatment phase was reduced stepwise by one step every week to the final dose level of paroxetine 20 mg/day as part of a taper phase.
Period: 4-Week Run-in Phase
Arm/Group | Placebo | Paroxetine 20-50 mg/Day
Started | 5 | 0
Completed | 3 | 0
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol-defined stopping criteria | 1 | 0
Period: 12-Week Treatment Phase
Arm/Group | Placebo | Paroxetine 20-50 mg/Day
Started | 1 | 2
Completed | 1 | 1
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Paroxetine 20-50 mg/Day | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Customized [Number; unit: participants]
  39 years old | 1 | 0 | 1
  43 years old | 0 | 1 | 1
  48 years old | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 1 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Asian-Japanese Heritage | 1 | 2 | 3
The number of participants with an MVA(Motor Vehicle Accident) of a particular duration [Number; unit: participants] — The number of participants who experienced a MVA of various durations with severe or potentially severe physical injury more than 3 months ago
  participants
    23 weeks | 0 | 1 | 1
    25 weeks | 0 | 1 | 1
    54 weeks | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Indicated Change From Baseline in CAPS-SX (Clinician-Administered Post Traumatic Stress Disorder (PTSD) Scale One Week Symptom Status Version) Total Score at Week 12
Description: The Clinical-Administered PTSD Scale (CAPS) is a structured interview for assessing PTSD diagnostic status and symptom severity. The CAPS assesses both the frequency and intensity of individual PTSD symptoms on separate five-point (0-4) rating scales, and these ratings can be summed to create a nine-point (0-8) severity score for each symptom. The total CAPS score can range from 0 to 136, with a higher value indicating increased severity. A minus value for change from baseline indicates an improvement of symptom severity.
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS): All participants who received at least one dose of study medication for the treatment phase and had at least one post-baseline efficacy assessment. Participants who failed to satisfy major entry criteria measured prior to randomization (e.g., participant with disease other than PTSD) were excluded.
Measure: Number; unit: participants
Arm/Group | Placebo | Paroxetine 20-50 mg/Day
Number analyzed (Participants) | 1 | 1
participants
  Change from baseline in CAPS-SX=+4 | 0 | 1
  Change from baseline in CAPS-SX=-27 | 1 | 0

2. Secondary Outcome: Number of Participants With the Indicated Week 0 and Week 12 Z-scores for Regional Blood Flow Using Functional Magnetic Resonance Imaging (fMRI) in the Left Amygdala (LA), Right Amygdala (RA), and the Medial Prefrontal Cortex (MPFC)
Description: Change in regional blood flow (rCBF) measured by fMRI represents altered neuronal responses in PTSD patients and is considered to be the biomarker for treatment response. fMRI measures are provided as blood oxygeneration level-dependent (BOLD) signals (z-score). To trigger neuronal activation, 2 visual stimuli were used: MVA-task (consisting of MVA-related and unpleasant pictures) and face-task (consisting of a variety of facial expressions [e.g., neutral, happy, fear]). Week 0 and 12 rCBF data from 1 participant were invalid (involuntary movement in the fMRI machine); no analysis was done.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Paroxetine 20-50 mg/Day
Number analyzed (Participants) | 1 | 2
participants
  LA: Week 0, MVA task, z-score of 6569 | 0 | 1
  LA: Week 0, MVA task, z-score of 2639 | 1 | 0
  LA: Week 0, face task, z-score of 5355 | 0 | 1
  LA: Week 0, face task, z-score of 2503 | 1 | 0
  LA: Week 12, MVA task, z-score of 2843 | 1 | 0
  LA: Week 12, face task, z-score of 2054 | 1 | 0
  RA: Week 0, MVA task, z-score of 6310 | 0 | 1
  RA: Week 0, MVA task, z-score of 2549 | 1 | 0
  RA: Week 0, face task, z-score of 4082 | 0 | 1
  RA: Week 0, face task, z-score of 3339 | 1 | 0
  RA: Week 12, MVA task, z-score of 2217 | 1 | 0
  RA: Week 12, face task, z-score of 2669 | 1 | 0
  MPFC: Week 0, MVA task, z-score of 10652 | 0 | 1
  MPFC: Week 0, MVA task, z-score of 3072 | 1 | 0
  MPFC: Week 0, face task, z-score of 6162 | 0 | 1
  MPFC: Week 0, face task, z-score of 5718 | 1 | 0
  MPFC: Week 12, MVA task, z-score of 9083 | 1 | 0
  MPFC: Week 12, MVA task, z-score of 3309 | 1 | 0

3. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in CAPS-SX (Clinician-Administered Post Traumatic Stress Disorder [PTSD] Scale One Week Symptom Status Version) Total Score at Weeks 4 and 8
Description: as for outcome 1
Time Frame: Baseline and Weeks 4 and 8
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Paroxetine 20-50 mg/Day
Number analyzed (Participants) | 1 | 1
participants
  Change in CAPS-SX total score=+7, Week 4 | 0 | 1
  Change in CAPS-SX total score=-4, Week 4 | 1 | 0
  Change in CAPS-SX total score=+10, Week 8 | 0 | 1
  Change in CAPS-SX total score=-10, Week 8 | 1 | 0

4. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in CAPS-SX (Clinician-Administered Post Traumatic Stress Disorder [PTSD] Scale One Week Symptom Status Version) Relating Re-experiencing at Weeks 4, 8, and 12
Description: as for outcome 1
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Paroxetine 20-50 mg/Day
Number analyzed (Participants) | 1 | 1
participants
  Change in CAPS-SX=+7, Week 4 | 0 | 1
  Change in CAPS-SX=-1, Week 4 | 1 | 0
  Change in CAPS-SX=+5, Week 8 | 0 | 1
  Change in CAPS-SX=-2, Week 8 | 1 | 0
  Change in CAPS-SX=+6, Week 12 | 0 | 1
  Change in CAPS-SX=-13, Week 12 | 1 | 0

5. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in CAPS-SX (Clinician-Administered Post Traumatic Stress Disorder [PTSD] Scale One Week Symptom Status Version) Relating Avoidance and Numbing at Weeks 4, 8, and 12
Description: as for outcome 1
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Paroxetine 20-50 mg/Day
Number analyzed (Participants) | 1 | 1
participants
  Change in CAPS-SX=0, Week 4 | 0 | 1
  Change in CAPS-SX=+1, Week 4 | 1 | 0
  Change in CAPS-SX=-3, Week 8 | 0 | 1
  Change in CAPS-SX=0, Week 8 | 1 | 0
  Change in CAPS-SX=-1, Week 12 | 0 | 1
  Change in CAPS-SX=-5, Week 12 | 1 | 0

6. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in CAPS-SX (Clinician-Administered Post Traumatic Stress Disorder [PTSD] Scale One Week Symptom Status Version) Relating Increased Arousal Symptom at Weeks 4, 8, and 12
Description: as for outcome 1
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Paroxetine 20-50 mg/Day
Number analyzed (Participants) | 1 | 1
participants
  Change in CAPS-SX=0, Week 4 | 0 | 1
  Change in CAPS-SX=-4, Week 4 | 1 | 0
  Change in CAPS-SX=+8, Week 8 | 0 | 1
  Change in CAPS-SX=-8, Week 8 | 1 | 0
  Change in CAPS-SX=-1, Week 12 | 0 | 1
  Change in CAPS-SX=-9, Week 12 | 1 | 0

7. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in CGI (Clinical Global Impression) Severity of Illness Scores at Weeks 2, 4, 6, 8, 10, and 12
Description: The participant's status was assessed using the following 8-point scale: 0, Not assessed; 1, Normal, not at all ill; 2, Borderline mentally ill; 3, Mildly ill; 4, Moderately ill; 5, Markedly ill; 6, Severely ill; 7, Among the most extremely ill patients.
Time Frame: Baseline and Weeks 2, 4, 6, 8, 10, and 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Paroxetine 20-50 mg/Day
Number analyzed (Participants) | 1 | 1
participants
  Change in CGI Severity of Illness=0, Week 2 | 1 | 0
  Change in CGI Severity of Illness=-1, Week 2 | 0 | 1
  Change in CGI Severity of Illness=0, Week 4 | 1 | 1
  Change in CGI Severity of Illness=0, Week 6 | 1 | 1
  Change in CGI Severity of Illness=0, Week 8 | 1 | 1
  Change in CGI Severity of Illness=0, Week 10 | 1 | 1
  Change in CGI Severity of Illness=0, Week 12 | 1 | 1

8. Secondary Outcome: Number of Participants With a Clinical Global Impression (CGI) Global Improvement of 4 at Week 12
Description: The participant's status was assessed using the following 8-point scale: 0, Not assessed; 1,Very much improved; 2, Much Improved; 3, Minimally improved; 4, No change; 5, Minimally worse; 6, Much worse; 7, Very much worse.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Paroxetine 20-50 mg/Day
Number analyzed (Participants) | 1 | 1
participants | 1 | 1

ADVERSE EVENTS:
Arm/Group | Placebo | Paroxetine 20-50 mg/Day
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1) | Paroxetine 20-50 mg/Day (N=2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Alanine aminotransferase increased (Hepatobiliary disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gamma-glutamyltransferase increased (Hepatobiliary disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Muscle tightness (Psychiatric disorders) | 1 | 0
Chorioretinopathy (Eye disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.